CLINICAL TRIAL: NCT06548425
Title: Effectiveness of Smartphone Based Tele-rehabilitation on Cardiovascular Functional Capacity and Sleep Quality Among Coronary Heart Disease Patients.
Brief Title: Smartphone Based Tele-rehabilitation on Functional Capacity and Sleep Quality Among Coronary Heart Disease Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/01890 Hassan
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Phone Based Cardiac Telerehabilitation (Experimental)
  Interventions: Other: Smart Phone Based Cardiac Telerehabilitation
- Center based cardiac Rehabilitation (Active Comparator)
  Interventions: Other: Center based cardiac Rehabilitation

INTERVENTIONS:
Other: Smart Phone Based Cardiac Telerehabilitation — Smart Phone Based Cardiac Telerehabilitation
  Frequency:3 sessions per week for 8 weeks Intensity: 40-60 % THR and modified borg scale 9 (very light- 13 (somewhat hard) Time: Approx. 30 Min Type: Aerobic & strength Exercises
  Arms: Smart Phone Based Cardiac Telerehabilitation
Other: Center based cardiac Rehabilitation — Center based cardiac Rehabilitation
  Frequency:3 sessions per week for 8 weeks Intensity: 40-60% THR and modified borg scale 9 (very light- 13 (somewhat hard)
  Time: Approx. 30 Min Type: Aerobic & strength Exercises
  Arms: Center based cardiac Rehabilitation

SUMMARY:
To determine the effectiveness of smartphone based tele-rehabilitation on functional capacity and sleep quality among coronary heart disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Both Male & Female
* Age 20-69 years
* Participants should have a documented diagnosis of CAD, confirmed by a medical professional.
* Individuals with a history of myocardial infarction (heart attack), angina, or evidence of significant coronary artery stenosis.
* Stable CAD who are not experiencing acute coronary events, such as recent heart attacks or unstable angina.

Exclusion Criteria:

* Acute illness
* Uncontrolled hypertension
* Uncontrolled metabolic disease
* Bone fracture in the last 6 months
* Neurological diseases that limit the ability to ambulate or stand from a chair
* MSK disease
* Severe cardiovascular complications such as heart failure with reduced ejection fraction, severe arrhythmias.
* Patients with unstable conditions or cardiac episodes.
* Ejection fraction < 40%

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 8 week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The PSQI has a high test-retest reliability and a good validity for patients with cardiac patients. Changes from the baseline will be measured.
Duke Activity Status Index | 8 week
  The Duke Activity Status Index (DASI) is an assessment tool used to evaluate the functional capacity of patients with cardiovascular disease (CVD), such as coronary artery disease, myocardial infarction, and heart failure. In clinical practice, DASI can be used to assess the effects of medical treatments and cardiac rehabilitation as well. Positive responses are summed up to get a total score, which ranges from 0 to 58.2. Higher scores would indicate a higher functional capacity. Changes from the baseline will be measured.
6 Minute walk test | 8 week
  six-minute walk test as a measure of functional status or fitness Before you begin to walk, the researchers will take a participant's blood pressure, pulse, and oxygen saturation using a pulse oximeter. Participants will get the instructions below. For six minutes, the contestants will walk as far as they can. to a chair or cone at your usual speed, then turn around. and will keep going back and forth for another six minutes. Distance will be measured in meters. Changes from the baseline will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Yusra Rehabilitation Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No